CLINICAL TRIAL: NCT02919384
Title: Evaluation of the Impact of Reduced Oxygen Concentration on Embryonic Development
Acronym: LO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol RMA-2016-02
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Infertility
Keywords: Embryonic development; blastocyst stage
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2% oxygen concentration in the incubator (Experimental): At the time that embryos are changed from "cleavage stage media" to "blastocyst stage media" on day 3 of development, half of a given patient's embryos will randomly be placed in an incubator set at 2% oxygen concentration. The splitting of the embryos will be done under low magnification such that the embryologist will have no ability to bias allocation of embryos to 2% or 5% oxygen based on embryo morphology on day 3. The embryos will remain in this incubator until their developmental assessments on day 5 and 6.
  Interventions: Other: 2% oxygen concentration in the incubator
- Control (No Intervention): Embryos in this arm will be cultured at 5% oxygen (current standard of care) from day 3 until blastocyst developmental assessment.

INTERVENTIONS:
Other: 2% oxygen concentration in the incubator — At the time that embryos are changed from "cleavage stage media" to "blastocyst stage media" on day 3 of development, half of a given patient's embryos will randomly be placed in an incubator set at 2% oxygen concentration. The splitting of the embryos will be done under low magnification such that the embryologist will have no ability to bias allocation of embryos to 2% or 5% oxygen based on embryo morphology on day 3. The embryos will remain in this incubator until their developmental assessments on day 5 and 6.
  Arms: 2% oxygen concentration in the incubator

SUMMARY:
During this study, patients will undergo a routine in vitro fertilization cycle as they would otherwise if not participating in the study. After eggs have been fertilized they will be cultured as usual until day 3 of embryo development. On day 3 of development, the embryologist will randomize half of the embryos to be cultured in 2% oxygen concentration and the other half at 5%, which is currently the standard of care. All other embryological care procedures will remain the same. On day 5 or 6 of embryo development, the embryos will be evaluated and each blastocyst stage embryo will be recorded. The primary outcome will be the blastulation rate (or percentage of embryos that reach the blastocyst stage).

DETAILED DESCRIPTION:
Significant progress has been made in characterizing the optimal environment for a developing embryo in culture. These efforts have been based on the premise that clinical embryo culture should mimic the in vivo environment. To this end, investigators have gone to great lengths to recreate every aspect of the natural setting to which the early embryo is exposed. This focused approach has led to significant modifications of the embryo culture system in the modern in vitro fertilization (IVF) lab and ultimately to improvements in pregnancy rates.

One area that has been subject to significant scrutiny is the relationship between incubator oxygen concentration and early embryonic development. Oxygen plays a central role in embryonic metabolism. The mechanism governing its utilization is dependent on the stage of embryonic development. During the first 3 days of development, oxygen reaches the embryo via passive diffusion and its concentration gradient is regulated by oxygen consumption during oxidative phosphorylation. Inefficiencies in this process - due to compromised integrity of the inner mitochondrial membrane or alterations in substrate availability - can result in excessive production of harmful reactive oxygen species which can cause significant damage to cellular machinery and ultimately lead to embryonic arrest.

The concentration of oxygen that the embryo in culture is exposed to can also impact this delicately balanced system and alter the metabolic health of an embryo. Historically, atmospheric oxygen concentration (approximately 20%) was exclusively used in human IVF laboratories for embryo culture. However, multiple investigations subsequently found that the physiologic concentration of oxygen within the female reproductive tract is well below atmospheric levels, being consistently measured at <10%. These observations led to multiple trials comparing atmospheric oxygen concentrations to 5% oxygen in embryo culture. These studies demonstrated significant perturbations in gene expression, protein secretion, and suboptimal utilization of amino acids and carbohydrates in embryos cultured in atmospheric oxygen. The same comparisons were made in clinical IVF studies and demonstrated that embryos cultured in 5% oxygen consistently resulted in an increase in clinical pregnancy rate and live birth rate. A meta-analysis of this topic suggested that a clinic with a baseline live birth rate of 30% could expect an improvement as great as 13% when culturing embryos at 5% O2.

As a result of these compelling data, most modern IVF programs now exclusively culture embryos at 5% oxygen concentration. However, some have proposed that the oxygen concentration to which the embryo is exposed after day 3 of development is actually lower than 5%. These data originate from the idea that the embryo crosses the utero-tubal junction on day 3 of development in vivo. Multiple studies have demonstrated that the oxygen concentration in the uterus is actually lower than that in the fallopian tube at approximately 2%. Thus, the most physiologic embryo culture system would culture embryos in 5% oxygen until day 3 and then decrease the oxygen concentration to 2% until transfer or cryopreservation on day 5 or 6.

A change in the optimal oxygen concentration for an embryo on day 3 would fit with a general shift in metabolic requirements of embryos seen at this stage of development. Activation of the embryonic genome occurs on day 3 which prompts a significant increase in biosynthetic activity. The metabolic behavior of embryos also shifts substantially during this time. The embryo changes its metabolic strategy from oxidative phosphorylation to glucose based metabolism in the form of the aerobic glycolysis and the citric acid cycle. During this process, termed compaction, embryos exhibit greatly increased oxygen consumption.

The physiologic environment of the female reproductive tract tends to mirror the metabolic needs of the developing preimplantation embryo. As the embryo shifts its metabolic strategy after compaction and upon entering the uterus, it is certainly possible that a reduced oxygen concentration in the uterus may best support the energy producing mechanisms of this stage in embryonic development. Recapitulating this environment in culture may enhance embryonic development and long term health of pregnancies resulting from IVF.

In fact a recent pilot study, using embryos donated to research demonstrated improved embryo development when embryos were cultured in 2% oxygen after day 3 of development compared to 5% (Kaser et al.)

Purpose of Proposed Study This study seeks to compare laboratory outcomes of embryos cultured at 2% oxygen concentration and 5% oxygen concentration after compaction. The primary outcome under study will be the proportion of day 3 embryos that are ongoing at the blastocyst stage (known throughout the rest of this document as blastulation rate).

A. Location of Study:

Patients will be recruited at both participating clinical centers. Oocyte retrieval, embryology, embryo biopsy, and embryo transfer will occur at the clinical facilities of Reproductive Medicine Associates of New Jersey. All genetic diagnostics will occur at the Foundation for Embryonic Competence (FEC).

B. Study Population:

Infertile couples attempting conception through in vitro fertilization. 60 couples will be enrolled in the study (see sample size calculation below).

STUDY PROCEDURES Experimental Design

The purpose of the study is to evaluate the embryological impact of 2% oxygen versus 5% concentrations in embryo culture after day 3 of development. As such, the study related procedures begin only after a patient's embryos reach day 3 of development.

The experimental design for this study is as follows: (Figure 1)

1. All care including oocyte retrieval, fertilization by ICSI, and cleavage stage culture (days 0, 1, and 2) will be completely per routine.
2. It is standard protocol in our laboratory to remove embryos from the incubator on day 3 to 1) perform assisted hatching and 2) change embryos from cleavage stage media to blastocyst media
3. At time of assisted hatching, two 5-well extended culture dishes will be brought to the isolette where changeover into extended culture will take place. The configuration of this 5-well dish is as follows. One mL of blastocyst media is placed in the center well of the 5-well dish. This well is only used for washing of cleavage stage embryos prior to placement into blastocyst media drops. The outer four wells contain small drops for ongoing blastocyst culture.

   As part of the study, once assisted hatching is complete, all embryos will be placed into the center well and mixed in the 1 mL of blastocyst media. At low power magnification and with no ability to perform day 3 grading, half of the embryos will be placed into the outer drops in one 5-well dish and half will be placed in the outer drops of the other 5-well dish. These two dishes will then be separated to the left and right side of the isolette. An embryologist, will then open a sequentially numbered, opaque sealed envelope from the box marked "oxygen randomization." The piece of paper in this envelope will direct the embryologist to place the 5-well dish on the left side of the isolette to either the 2 or 5% oxygen concentration incubator. The 5-well dish on the right side of the incubator will go to the opposite condition.
4. The number of ongoing day 3 embryos in each condition will then be recorded and given to data assessors.
5. Embryos will not be examined or manipulated at all until day 5 of development as per routine protocol.
6. On day 5 or 6 of embryo development, the embryos will be evaluated and the number of ongoing blastocysts will be recorded for embryos cultured in each condition.
7. All ongoing embryos will then undergo a trophectoderm biopsy using the standardized technique according to standard laboratory protocol without regard to study. Embryos will then be cryopreserved to allow for results from comprehensive chromosomal screening to be available and to optimize embryonic-endometrial synchrony, as per standard protocol.
8. Further decisions regarding the number of euploid embryos to transfer will be up to the patient. Data will be collected regarding pregnancy outcomes according to the culture conditions that a transferred embryo was exposed. However, all of this information will be analyzed as secondary outcomes.
9. Pregnancy testing and follow up will not be altered.

RANDOMIZATION SCHEMA

Simple randomization will be performed independently at the study site (RMANJ). A random number sequence will be generated by random.org. Odd numbers will be assigned to A intervention (2%) oxygen and even numbers will be assigned to B intervention (5%). Pieces of paper containing the letter dictated by random number sequence will be placed into a box of sequentially numbered, opaque sealed envelopes labelled "oxygen randomization."

As noted above, on day 3, after placing half of the embryos into one 5-well dish and half of the embryos into another 5-well dish, the embryologist will separate those dishes to the left and right hand side of the incubator. The embryologist, will then open a sequentially numbered, opaque sealed envelope from this box marked "oxygen randomization." The piece of paper in this envelope will direct the embryologist to place the 5-well dish on the left side of the isolette to either the 2 or 5% oxygen concentration incubator. The 5-well dish on the right side of the incubator will go to the opposite condition.

In the case of an odd number of embryos, the extra embryo will always be placed in the left handed 5-well dish. The numbers are anticipated to even out as the left sided dish has an equal chance of randomization to 2 or 5% oxygen concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years and seeking IVF with aneuploidy screening, which is our current recommendation regardless of study participation
2. Anti-mullerian hormone level (AMH) > 1.0 pmol/L (an assessment of ovarian reserve)
3. Must have at least two surviving embryos on day 3 of development
4. Male partner with >100,000 total motile spermatozoa per ejaculate (donor sperm acceptable)
5. Body Mass Index < 35

Exclusion Criteria:

1. Diagnosis of endometrial insufficiency, as defined by prior cycle with maximal endometrial thickness <6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), or persistent endometrial fluid
2. Use of oocyte donation
3. Use of gestational carrier
4. Use of sperm obtained via surgical procedure
5. Presence of hydrosalpinges that communicate with endometrial cavity
6. Single gene disorders, chromosomal translocations or any other disorders requiring more detailed embryo genetic analysis
7. Couples seeking gender selection for family balancing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Blastulation Rate (number of embryos meeting criteria for biopsy and/cryopreservation divided by number of embryos randomized on day 3 to either the experimental or control arm) | 6 days of embryonic development in the laboratory
  On day 5 and day 6, all embryos are examined under the microscope to see if they 1) meet developmental criteria for embryo biopsy (for chromosomal evaluation) and cryopreservation (since all embryos in this program are cryopreserved while awaiting results from chromosome assessment), or 2) arrest development in the laboratory.

SECONDARY OUTCOMES:
Clinical Pregnancy rate | 2 months
  After embryos are cryopreserved, embryos with the proper number of chromosomes (so called euploid embryos) will be available for transfer to the uterus (as is standard protocol in our center). Clinical pregnancy rate will be defined by the presence of a gestational sac on ultrasound in the embryo transfer cycle.

OTHER OUTCOMES:
Live birth rate | 10 months
  Delivery of an alive baby will be the criteria for live birth rate assessment

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Morin, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer B, Bavister BD. Oxygen tension in the oviduct and uterus of rhesus monkeys, hamsters and rabbits. J Reprod Fertil. 1993 Nov;99(2):673-9. doi: 10.1530/jrf.0.0990673. PMID 8107053
- [Background] Bontekoe S, Mantikou E, van Wely M, Seshadri S, Repping S, Mastenbroek S. Low oxygen concentrations for embryo culture in assisted reproductive technologies. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008950. doi: 10.1002/14651858.CD008950.pub2. PMID 22786519
- [Background] Gardner DK, Wale PL. Analysis of metabolism to select viable human embryos for transfer. Fertil Steril. 2013 Mar 15;99(4):1062-72. doi: 10.1016/j.fertnstert.2012.12.004. Epub 2013 Jan 8. PMID 23312219
- [Background] Meintjes M, Chantilis SJ, Douglas JD, Rodriguez AJ, Guerami AR, Bookout DM, Barnett BD, Madden JD. A controlled randomized trial evaluating the effect of lowered incubator oxygen tension on live births in a predominantly blastocyst transfer program. Hum Reprod. 2009 Feb;24(2):300-7. doi: 10.1093/humrep/den368. Epub 2008 Oct 16. PMID 18927130